CLINICAL TRIAL: NCT03421795
Title: Let's Talk About Pain: A Randomized Controlled Trial Testing the Effectiveness of a Pain Assessment and Management Training Program for Respite Workers Supporting Children With Intellectual and Developmental Disabilities
Brief Title: Effectiveness of a Pain Assessment and Management Program for Respite Workers Supporting Children With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Society of Pediatric Psychology (Unknown); Western University (Other)
Responsible Party: Principal Investigator, Meghan McMurtry, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB16-12-696
Record Dates: First submitted 2017-12-12; First posted 2018-02-05 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Pain
Keywords: pain assessment/management; developmental disabilities; children; education; respite workers
MeSH Terms: conditions — Pain; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: This is a multi-centre clustered parallel RCT with an intervention group (pain training) and control group (control training about family centered care, with an option to receive pain training after follow-up).
Masking Description: Organizations will not be made explicitly aware of whether they have been allocated as part of the control or experimental conditions. Organizations will be told, however, that if they are not assigned to the experimental group, they will be given the option to also have an additional training about pain in children with DD at the end of the study. They will also know about the topics of both training programs and the purpose of the study. Participants will only be told that the purpose of the study is to learn about the impact that training programs can have on respite workers' knowledge about caring for children with DD. However, given some of the information in the consent form (e.g., study title is "Let's Talk about Pain"), it is likely that the treatment condition is clear to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Let's Talk About Pain Training (Experimental): Participants complete pre-, post- and follow-up measures, and receive a pain training program. The pain assessment and management training will be based on a training previously developed and piloted by Genik et al. (2017). The training will be facilitated by the same researcher (L.G.) throughout the study.
  Interventions: Other: Let's Talk About Pain Training
- Family Centered Care Training (Sham Comparator): Participants complete all of the same measures as those in the intervention, but receive a training about family centered care. This training will be facilitated by Andrea Cross (PhD Candidate) from CanChild and will be related to the F-words of childhood disability (function, family, fitness, fun, friends, future; Rosenbaum & Gorter, 2012) .
  Interventions: Other: Family Centered Care Training

INTERVENTIONS:
Other: Let's Talk About Pain Training — See arm/group descriptions.
  Arms: Let's Talk About Pain Training
Other: Family Centered Care Training — See arm/group descriptions.
  Arms: Family Centered Care Training

SUMMARY:
This study investigates the impact of pain training delivery for respite care providers who support children with developmental disabilities on (a) pain assessment and management-related knowledge, (b) participant self-rated perceptions of the feasibility, confidence and skill in pain assessment and management, and (c) strategy use. Half of the participants will receive the pain training, while half will receive the training about family-centered care, and be offered the pain training after completion of the follow-up.

DETAILED DESCRIPTION:
Background Information: Everyday pain is common in children with intellectual/developmental disabilities (I/DD). Inadequately managed pain in this population is a common problem, and this is likely due to these children's inability to communicate pain effectively. Unfortunately, many of these children are unable to accurately self-report or effectively communicate the pain experience. Thus, caregivers are often responsible for assessing their pain. Research has focused on professionals and parents, but it is also common for children with I/DD to receive care from others including respite workers. The investigators recently found a difference between pain beliefs held by respite workers and individuals with little to no experience with this population. Specifically, respite workers believed that a significantly larger percentage of children with severe I/DD sensed less pain than typically developing children. This is contrary to research suggesting that children with I/DD have similar pain perception but communicate it differently (e.g., through idiosyncratic behaviours). Thus, it is possible that respite workers miss critical cues when children with I/DD are in pain. As such, the investigators have developed and successfully piloted a pain training program targeted to respite workers who support children with I/DD. This program demonstrated initial success in improving respite workers' pain-related knowledge, as well as their perceptions of the feasibility of and their own confidence and skill in pain assessment and management with this population of children.

Within a randomized control trial, the objectives of this study are to further test the effectiveness of the Let's Talk About Pain respite worker training program on respite workers' (a) pain-related knowledge, (b) self-rated perceptions of the feasibility of and their own confidence and skill in pain assessment and management, and (c) use of pain assessment and management strategies specific to children with I/DD in respite settings. Participants will complete questionnaires immediately before and after provision of a pain training (or control training). Approximately one month after the training, participants will complete these questionnaires for a third time and participate in a focus group regarding their pain assessment and management strategy use.

The long term objectives of this line of research are to: 1) increase pain assessment and management abilities of respite workers, and, consequently, 2) decrease levels of suffering and ill-managed pain in children with I/DD.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Proficient in the English language
* Active respite worker who provides respite care to children (age 0 - 18) with developmental disabilities

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Within intervention group change from baseline in scores on Questionnaire for Understanding Pain in Individuals with Intellectual and Developmental Disabilities - Revised | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Pain-related knowledge assessment
Within intervention group change (i.e., maintenance) from post in scores on Questionnaire for Understanding Pain in Individuals with Intellectual and Developmental Disabilities - Revised | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Pain-related knowledge assessment
Between group difference in scores on Questionnaire for Understanding Pain in Individuals with Intellectual and Developmental Disabilities - Revised | Post (within 30 minutes after completion of training)
  Pain-related knowledge assessment
Between group difference in scores on Questionnaire for Understanding Pain in Individuals with Intellectual and Developmental Disabilities - Revised | Follow-Up (approximately one month after training)
  Pain-related knowledge assessment

SECONDARY OUTCOMES:
Between group difference in ratings of the feasibility of pain assessment | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain assessment; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Between group difference in ratings of the feasibility of pain assessment | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain assessment; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Between group difference ratings of the feasibility of pain management | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain management; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Between group difference ratings of the feasibility of pain management | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain management; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Between group difference ratings of perceived confidence in pain assessment abilities | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain assessment abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Between group difference ratings of perceived confidence in pain assessment abilities | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain assessment abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Between group difference ratings of perceived confidence in pain management abilities | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain management abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Between group difference ratings of perceived confidence in pain management abilities | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain management abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Between group difference ratings of perceived skill in pain assessment | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain assessment; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Between group difference ratings of perceived skill in pain assessment | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain assessment; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Between group difference ratings of perceived skill in pain management | Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain management; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Between group difference ratings of perceived skill in pain management | Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain management; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of the feasibility of pain assessment | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain assessment; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of the feasibility of pain management | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain management; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of perceived confidence in pain assessment | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain assessment abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of perceived confidence in pain management | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain management abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of perceived skill in pain assessment | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain assessment; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Within intervention group change from baseline in ratings of perceived skill in pain management | Baseline (within 30 minutes prior to start of training), Post (within 30 minutes after completion of training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain management; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of the feasibility of pain assessment | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain assessment; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of the feasibility of pain management | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of the feasibility of pain management; 0 (Not feasible at all) - 10 (highly/extremely feasible) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of perceived confidence in pain assessment | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain assessment abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of perceived confidence in pain management | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own confidence in their pain management abilities; 0 (Not confident at all) - 10 (highly/extremely confident) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of perceived skill in pain assessment | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain assessment; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.
Within intervention group change (i.e., maintenance) from post in ratings of perceived skill in pain management | Post (within 30 minutes after completion of training), Follow-Up (approximately one month after training)
  Researcher generated scale measuring participants' perceptions of their own skill in pain management; 0 (Not skilled at all) - 10 (highly/extremely skilled) Likert Scale. Higher scores are better.

OTHER OUTCOMES:
Between group difference in use of evidence-based pain assessment and management strategies as indicated on a researcher-generated questionnaire and in focus groups | Follow-Up (approximately one month after training)
  Assessment of use of evidence-based pain assessment and management strategies (researcher generated questionnaire with open-ended responses and focus groups)
Within intervention group change from baseline in use of evidence-based pain assessment and management strategies as indicated on a researcher-generated questionnaire | Baseline (within 30 minutes prior to start of training), Follow-Up (approximately one month after training)
  Assessment of use of evidence-based pain assessment and management strategies (researcher generated questionnaire)
Within intervention group descriptive ratings of training | Post (within 30 minutes after completion of training)
  Assessment of training program endorsement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubois A, Capdevila X, Bringuier S, Pry R. Pain expression in children with an intellectual disability. Eur J Pain. 2010 Jul;14(6):654-60. doi: 10.1016/j.ejpain.2009.10.013. Epub 2009 Dec 5. PMID 19963417
- [Background] Twycross A, Williams A. Establishing the validity and reliability of a pediatric pain knowledge and attitudes questionnaire. Pain Manag Nurs. 2013 Sep;14(3):e47-53. doi: 10.1016/j.pmn.2011.03.001. Epub 2011 Apr 17. PMID 23972870
- [Background] Chen-Lim ML, Zarnowsky C, Green R, Shaffer S, Holtzer B, Ely E. Optimizing the assessment of pain in children who are cognitively impaired through the quality improvement process. J Pediatr Nurs. 2012 Dec;27(6):750-9. doi: 10.1016/j.pedn.2012.03.023. Epub 2012 Apr 10. PMID 22497741
- [Background] Genik LM, McMurtry CM, Breau LM. Caring for children with intellectual disabilities part 1: Experience with the population, pain-related beliefs, and care decisions. Res Dev Disabil. 2017 Mar;62:197-208. doi: 10.1016/j.ridd.2017.01.020. Epub 2017 Feb 14. PMID 28208103
- [Background] Genik LM, McMurtry CM, Breau LM, Lewis SP, Freedman-Kalchman T. Pain in Children With Developmental Disabilities: Development and Preliminary Effectiveness of a Pain Training Workshop for Respite Workers. Clin J Pain. 2018 May;34(5):428-437. doi: 10.1097/AJP.0000000000000554. PMID 28877138
- [Background] Breau LM, MacLaren J, McGrath PJ, Camfield CS, Finley GA. Caregivers' beliefs regarding pain in children with cognitive impairment: relation between pain sensation and reaction increases with severity of impairment. Clin J Pain. 2003 Nov-Dec;19(6):335-44. doi: 10.1097/00002508-200311000-00001. PMID 14600533
- [Derived] Genik LM, McMurtry CM, Barata PC, Barney CC, Lewis SP. Study protocol for a multi-centre parallel two-group randomized controlled trial evaluating the effectiveness and impact of a pain assessment and management program for respite workers supporting children with disabilities. Paediatr Neonatal Pain. 2020 Apr 26;2(1):7-13. doi: 10.1002/pne2.12014. eCollection 2020 Mar. PMID 35547857